CLINICAL TRIAL: NCT03704467
Title: A Phase Ib Safety Run-in and Randomized Phase II, Open-label Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of M6620 in Combination With Avelumab and Carboplatin in Comparison to Standard of Care Therapy in Participants With PARPi-resistant Recurrent Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: Phase Ib/II Study of Carboplatin + M6620 + Avelumab in PARPi-resistant Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS201943_0029; 2018-001534-17 (EudraCT Number)
Record Dates: First submitted 2018-10-03; First posted 2018-10-12 (Actual); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Ovarian Cancer
Keywords: Avelumab; Carboplatin; Primary Peritoneal Cancer; Fallopian Tube Cancer; Platinum sensitive ovarian cancer; Deoxy ribonucleic acid (DNA)-damage response inhibition
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — avelumab; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part A: Carboplatin + M6620 + Avelumab (Experimental)
  Interventions: Drug: M6620; Drug: Avelumab; Drug: Carboplatin

INTERVENTIONS:
Drug: M6620 — Participants received 90 milligrams per square meter (mg/m^2) of M6620, intravenously (IV) on Day 2 of every 3 weeks (Q3W) cycle for a maximum of 6 cycles in combination treatment with carboplatin and avelumab on Day 1. The M6620 dose may be de-escalated to 60 mg/m^2, or 40 mg/m^2.
Drug: Avelumab — Participants received IV infusion of avelumab 1600 mg on Day 1 of each Q3W cycle for maximum of 6 cycles in combination treatment with carboplatin and M6620. Thereafter, avelumab 800 mg intravenously on Day 1 of every two weeks as a maintenance mono-therapy until progressive disease (PD), unacceptable toxicity, withdrawal of consent, or death.
Drug: Carboplatin — Participants received carboplatin area under the concentration-time curve 5 on Day 1 of each Q3W cycle for a maximum of 6 cycles in combination treatment with avelumab and M6620.

SUMMARY:
The study was to evaluate the efficacy and safety of avelumab in combination with M6620 + carboplatin in participants with PARPi-resistant, recurrent, platinum sensitive ovarian, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
The study was intended to be a phase Ib/II trial, but after completing Phase 1b and confirming the safe combination dose, the sponsor decided not to conduct Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Female participants with recurrent epithelial ovarian cancer who have disease progression following maintenance treatment with a PARPi as defined below:

  1. Participant must have histologically diagnosed epithelial ovarian, primary peritoneal, or fallopian tube cancer, with nonmucinous histology
  2. Participants must have completed at least 2 previous courses of platinum containing therapy (for example, carboplatin or cisplatin) and had documented response (complete response [CR] or partial response [PR]) to the last platinum-based treatment prior to treatment with a PARPi
  3. Participant has received the last dose of platinum-containing treatment at least 6 months prior to study enrollment
  4. Participant has documented disease progression (radiological) after at least 4 months of maintenance treatment with PARPi following a response to platinum-based chemotherapy.
* Confirmed breast cancer gene (BRCA) 1/2 mutation status or agree to its testing on samples collected in the study.
* Available formalin-fixed, paraffin-embedded (FFPE) tumor biopsies.
* Part A: Optional 2 paired on-treatment biopsies on Day 2 of Cycle 1 (first biopsy) and Day 2 of Cycle 1 or Cycle 2 (second biopsy) respectively, before and after M6620 administration, if assessed as feasible at low risk by the interventional radiologist.
* Part B: Histological tissue specimen (tissue block or 8 to 10 unstained slides) must be available. An archival tumor biopsy is acceptable if obtained after the last progression on PARPi treatment and is less than 4 months old. Otherwise, participants must be willing to undergo mandatory biopsy during the Screening Period to obtain sufficient tissue for histological assessment. Participants need to have an attempted biopsy. However, participants who have measurable disease documented by a radiologist as not feasible or safe to be biopsied are eligible to enter the study
* Measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Treatment with a nonpermitted drug/intervention as listed below:

  1. Concurrent anticancer treatment (e.g., cytoreductive therapy, radiotherapy, immune therapy, cytokine therapy, monoclonal antibody, or targeted small molecule therapy) or any study intervention within 4 weeks prior to start of study intervention, or not recovered from AEs related to such therapies
  2. History of prior dose reductions or dose interruptions while receiving cisplatin or carboplatin due to toxicity from the platinum or intolerance to either agent, unless discussed with and approved by the Sponsor Medical Monitor
  3. Prior treatment with a PD-1/PD-L1 targeting agent
* Current use of the following medications at the time of enrollment:

  1. Immunotherapy or immunosuppressive drugs at the time of enrollment (for example (e.g.,) chemotherapy or systemic corticosteroids) EXCEPT for (a) intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra articular injection), (b) systemic corticosteroids at physiologic doses less than or equals to (≤) 10 milligram per day (mg/day) of prednisone or equivalent, (c) steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
  2. Growth factors EXCEPT where indicated for treatment of study intervention related myelosuppression and for prophylaxis of repeat myelosuppression after initial occurrence
  3. Herbal remedies with immunostimulating properties (e.g., mistletoe extract) or known to potentially interfere with major organ function (e.g., hypericin)
  4. Other DNA damage repair inhibitors (except PARPi) (e.g., inhibitors of ATR, ataxia telangiectasia mutated [ATM] kinase, DNA-dependent protein kinase [DNA-PK], or Wee kinases).
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (13):
- United States (7):
  - Marin Cancer Care, Inc., Greenbrae, California
  - The Stamford Hospital, Stamford, Connecticut
  - Covenant Health Care, Saginaw, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mount Sinai - PRIME, New York, New York
  - Peggy & Charles Stephenson Oklahoma Cancer Ctr, Oklahoma City, Oklahoma
  - Mary Crowley Cancer Research Centers, Dallas, Texas
- Belgium (3):
  - UZ Leuven, Leuven
  - CHU Sart Tilman, Liège
  - GZA Ziekenhuizen - Campus Sint-Augustinus, Wilrijk
- United Kingdom (3):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Royal Marsden Hospital, Sutton, Surrey
  - Royal Marsden Hospital, London

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201943_0029
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant signed informed consent: 04 Mar 2019, Last participant last visit: 06 Nov 2019.
Pre-assignment Details: This study was planned to be conducted in 2 parts; Part A was the safety run-in part and Part 2 was the randomized controlled part. However, after completing Part A and confirming the safe combination dose, the sponsor decided not to conduct Part B.
Groups:
- Part A: Carboplatin + M6620 + Avelumab: Participants received intravenous infusion of Carboplatin area under the concentration-time curve 5 on Day 1 in combination with 90 milligrams per square meter (mg/m^2) of M6620 on Day 2 and avelumab at an established dose of 1600 mg over 60 minutes on Day 1 for every 3 weeks cycle for a maximum of 6 cycles. Thereafter, avelumab 800 mg intravenously on Day 1 of every two weeks as a maintenance mono-therapy until progressive disease (PD), unacceptable toxicity, withdrawal of consent, or death.
Period: Overall Study
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of any study intervention.
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT: any death not clearly due to underlying disease/extraneous causes/Grade(Gr) >=3 nonhematologic/Gr>=4 hematologic toxicity that was probably/definitely related to any of study interventions, individually/combination that occurred during DLT observation period, except for any of following: Gr3 infusion-related reaction; Transient (<=6hr) Gr3 flu-like symptoms/fever, controlled with medical management; Transient (<=72hr) Gr3 fatigue, local reactions, headache, nausea/emesis; Gr3 diarrhea, skin toxicity, liver function test increase; Single laboratory values out of normal range and controlled with medical management; Tumor flare phenomenon: local pain, irritation/rash, localized at sites of known/suspected tumor; Neutropenia (Gr3/4) for <7 days not associated with any infection; Gr3 thrombocytopenia for <7 days without clinically significant bleeding and not requiring platelet transfusion; Symptomatic thyroid dysfunction manageable with treatment.
Time Frame: Up to 3 weeks
Population: DLT analysis set included all evaluable participants with data used for implementing the dose-escalation schedule. These participants received at least 1 study intervention administration of each avelumab, M6620, and/or chemotherapy in the DLT evaluation period or should have stopped treatment because of DLTs in the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Part A: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were defined as events that started or worsened after first dose of study intervention until 30 days after last dose. TEAEs included both serious and non-serious AEs. Treatment-related TEAE: reasonably related to the study intervention. The AE could medically (pharmacologically/clinically) be attributed to the study intervention under study in this clinical study protocol.
Time Frame: Time from first dose of study treatment up to 230 days
Population: Safety analysis set included all participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 3
Participants
  TEAEs | 3
  Treatment-Related TEAEs | 3

3. Secondary Outcome: Part A: Number of Participants With Confirmed Best Overall Response (BOR)
Description: Confirmed BOR according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and as assessed by an Investigator was defined as best response of any of the complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) recorded from the date of randomization until disease progression/ recurrence (taking the smallest measurement recorded since the start of treatment as reference). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. SD: Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions and unequivocal progression of non-target lesions. Number of participants with BOR in each category (CR, PR, SD, PD) were reported.
Time Frame: Time from first dose of study treatment up to 230 days
Population: Safety analysis set included all participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 3
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 1
  Progressive Disease | 2

4. Secondary Outcome: Part A: Progression-Free Survival (PFS)
Description: PFS according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and as assessed by an Investigator was defined as the time from date of randomization until date of the first observation of progressive disease (PD) or death due to any cause within 12 weeks of the last tumor assessment in the absence of documented PD, whichever occurs first. PD was defined as at least a 20% increase in the sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions and unequivocal progression of non-target lesions. Participant wise data reported for this outcome measure.
Time Frame: Time from first dose of study treatment up to 230 days
Population: Safety analysis set was used. No summary analysis was done as study was early discontinued as per Sponsor's decision and participant wise data was reported. Here, "Number Analyzed" signifies specific participant evaluated in the arm of this outcome measure.
Measure: Number; unit: months
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 3
months
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 1.9
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 2.1
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 6.1

5. Secondary Outcome: Part A: Duration of Response (DoR)
Description: DoR according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and as assessed by an Investigator was defined as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of objective progression of disease (PD) or death due to any cause whichever occurs first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions and unequivocal progression of non-target lesions. If a participant has not an event (PD or death), DoR was censored at the date of last adequate tumor assessment.
Time Frame: Time from first dose of study treatment up to 230 days
Population: Data could not be calculated as none of the participants showed objective response.
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Part A: Time to Progression (TTP)
Description: TTP according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and assessed by an Investigator was defined as the time from first dose of study intervention until progression disease (PD). PD was defined as at least a 20% increase in the sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions and unequivocal progression of non-target lesions. Participant wise data reported for this outcome measure.
Time Frame: Time from first dose of study treatment up to 230 days
Population: Safety analysis set was used. No summary analysis was done as study was early discontinued as per Sponsor's decision and participant wise data was reported. Here, "Overall Number of Participants Analyzed" = participants who were evaluable for this outcome measure and "number analyzed" = specific participants evaluated in the arm.
Measure: Number; unit: months
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 2
months
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 1.9
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 2.1

7. Secondary Outcome: Part A: Time to First Subsequent Therapy (TFST)
Description: The TFST was defined as the time from the date of randomization to the start date of the first subsequent anti-cancer therapy or death.
Time Frame: From date of randomization to the earliest date of first subsequent therapy or death, assessed up to 230 days
Population: Data could not be calculated since the date of first subsequent treatment was not recorded in the electronic case report form (eCRF) as per changes in planned analysis.
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) of M6620 and Avelumab
Description: Area under the plasma concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0, 1, 2, 3 and 6 hours post-dose on Day 2 Cycle 1; post-dose 47 hours on Day 4 Cycle 1; pre-dose and at 0 hour on Day 2 Cycle 2 (each Cycle is 21 days)
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M6620 and Avelumab
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: as for outcome 8
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Curve During a Dosing Interval (AUCtau)
Description: AUCtau was defined as area under the plasma concentration-time curve from time zero to the end of the dosing interval (tau). AUCtau was calculated using the mixed log linear trapezoidal rule.
Time Frame: as for outcome 8
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Part A: Terminal Rate Constant (Lambda z) of M6620 and Avelumab
Description: Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: as for outcome 8
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 0

12. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of M6620 and Avelumab
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 8
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 0

13. Secondary Outcome: Part A: Minimum Observed Plasma Concentration (Cmin) of M6620 and Avelumab
Description: Cmin was minimum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 8
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 0

14. Secondary Outcome: Part A: Time to Reach the Maximum Plasma Concentration (Tmax) of M6620 and Avelumab
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 8
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 0

15. Secondary Outcome: Part A: Apparent Terminal Half-life (t1/2) of M6620 and Avelumab
Description: t1/2 was the time measured for the concentration to decrease by one half. t1/2 was calculated by natural log 2 divided by Lambda z.
Time Frame: as for outcome 8
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Time from first dose of study treatment up to 230 days
Arm/Group | Part A: Carboplatin + M6620 + Avelumab
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Carboplatin + M6620 + Avelumab (N=3)
Pyelonephritis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Carboplatin + M6620 + Avelumab (N=3)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Fatigue (General disorders) | 2
Peripheral swelling (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Tooth infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Tooth fracture (Injury, poisoning and procedural complications) | 1
Blood urine present (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Bladder pain (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study was early discontinued and Part 2 (randomized controlled) was not conducted as per Sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT03704467/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT03704467/SAP_001.pdf